CLINICAL TRIAL: NCT07294820
Title: The Use of a Fully Digital Workflow in Immediate Implants With Immediate Restoration
Status: Recruiting | Type: Observational
Sponsor: Proed, Torino, Italy (Other)
Responsible Party: Principal Investigator, Daniele Cardaropoli, Prof Dr, Proed, Torino, Italy
Other Study IDs: 12.2025.IIPP.STR.IIS07/24
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Implant Dentistry
Keywords: oral implant placement; computer guided surgery; Immediata implant placement
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: oral implant — fully guided implant placement with a computer guided surgical stant

SUMMARY:
Study hypothesis The hypothesis is that a full-digital workflow for immediate implant placement with immediate restoration is able to provide at least the same outcomes as standard analog implant placement in the same clinical scenario (immediate placement with immediate loading), in terms of implant success and survival and marginal bone level stability. A VAS scale evaluation will be created to measure patients' aesthetic and overall satisfaction, as well the duration of the procedure will be measured.

Type of study Clinical

Study design Prospective, single-arm using BLC implants with full digital workflow. Patients treated within "Clinical and radiological evaluation of a novel implant design (Straumann BLX) in the esthetic zone: a prospective case series study" (IIS 43/17), published as "Cardaropoli D, Tamagnone L, Roffredo A, Demaria A. Clinical and radiological evaluation of a fully tapered implant with immediate placement in the aesthetic zone: a prospective case series study. Int J Periodontics Restorative Dent. 2022 Sep-Oct;42(5):631-637" will be used for comparison.

Study power N total: 24 Anticipated drop-out rate %: 15 Adequate power analysis and justification A power calculation before the study revealed that a sample size of 20 was necessary to detect a difference of 0.5 mm in the vertical position of the implant between planning and execution of 0.5 mm assuming a maximal standard deviation of 0.7 mm using a paired t test with 80% power and .05 level of significance.

Study intervention - test arm Study Device BLC Implant

Test treatment name Fully digital immediate placement/immediate restoration

Test Treatment description An immediate BLC implant inserted in post-extraction sites in the upper maxilla, from 15 to 25, with immediate restoration.

Primary outcome parameter Pink Esthetic Score (PES from 0 to 14), at 1 year Marginal Bone Level expressed in mm, at 1 year

Secondary outcome parameter PROMS - Patients' satisfaction using VAS scale, at day of surgery and at 1 year Duration of the procedure, at day of surgery Probing Depth (PD) and Bleeding on Probing (BoP) at 1 year

Materials and Methods Population and indication 24 adult systemically healthy patients requiring tooth extraction and single implant tooth replacement, from 1.5 to 2.5

Treatments In the case study phase, a 3D cone-beam radiograph and an intraoral scan are acquired. A computer guided surgical stent is produced from the virtual planning. By sharing the virtual planning, the laboratory designs and produces a temporary crown. On the day of surgery the tooth is extracted, the implant is inserted and the temporary is delivered. The final ceramic crown is delivered 3 months later. Follow-up will end 1 year after implant placement.

DETAILED DESCRIPTION:
Summary Immediate implant placement is a procedure that can have enormous benefits from using a fully digital workflow. The pre-surgical planning phase can be performed by combining cone-beam images with intraoral scanning. This matching allows you to pre-visualize the extraction of the tooth, making a careful assessment of the bone volume available in the post-extraction socket, and to plan the implant insertion according to the indications reported in the literature. A computer guided surgical stent can be printed "in office" from the plan. At the same time, the planning is exported to the cloud so that it can be viewed by the laboratory that will carry out the provisional crown. On the day of the surgery, with a minimally invasive procedure, after the extraction of the tooth and the insertion of the implant, the implanted temporary crown will be immediately delivered to the patient.

Background and rationale Immediate implant insertion is a treatment protocol that allows the insertion of an osseointegrated implant at the same time as tooth extraction. This procedure has high success rates, above 98%, but at the same time a high risk of biological and aesthetic complications. If possible, the delivery of an immediate temporary crown can improve the aesthetic result in terms of maintaining the original soft tissue profile. Planning the intervention becomes a fundamental point in the diagnostic-therapeutic path. It is essential to have three-dimensional radiographic information in order to evaluate the buccal bone plate, and the post-extractions socket. But it is also very important to have detailed information about the position and quality of the soft tissues. This information can be made available by cone-beam radiographic examination and intraoral digital scanning. The digital planning of the implant surgery can be shared with the laboratory which will design the temporary crown and produce it. On the day of surgery, thanks to the computer guided surgical stent, the implant can be inserted in the three-dimensional position as chosen and at the end of the session the temporary crown with its temporary abutment will be delivered. The fully digital workflow can create a minimally invasive, fast and precise treatment protocol, capable of pre-visualizing unfavorable anatomical conditions.

The outcome of this study will be compared with the results obtained from the recently completed clinical trial with similar design (Cardaropoli D, Tamagnone L, Roffredo A, Demaria A. Clinical and radiological evaluation of a fully tapered implant with immediate placement in the aesthetic zone: a prospective case series study. Int J Periodontics Restorative Dent. 2022 Sep-Oct;42(5):631-637.). In this study fully tapered implants with comparable design (BLX) have been placed in post-extraction sockets, from premolar to premolar in the maxilla, and immediately loaded. Marginal bone level (MBL) and probing depth (PD) have been evaluated up to a 12-month follow-up period. All implants osseointegrated achieving a success rate of 100%. Difference in MBL between time of placement and one year was 0.20 ± 0.04 mm, while PD at one year was 2.82±0.51. Data here reported support the use of a fully tapered implant for immediate placement and immediate loading, for single-tooth replacements in the aesthetic area.

Study hypothesis The hypothesis is that a full-digital workflow for immediate implant placement with immediate restoration is able to provide at least the same outcomes as standard analog implant placement in the same clinical scenario (immediate placement with immediate loading), in terms of implant success and survival and marginal bone level stability. A VAS scale evaluation will be created to measure patients' aesthetic and overall satisfaction, as well the duration of the procedure will be measured.

Type of study Clinical

Study design Prospective, single-arm using BLC implants with full digital workflow. Patients treated within "Clinical and radiological evaluation of a novel implant design (Straumann BLX) in the esthetic zone: a prospective case series study" (IIS 43/17), published as "Cardaropoli D, Tamagnone L, Roffredo A, Demaria A. Clinical and radiological evaluation of a fully tapered implant with immediate placement in the aesthetic zone: a prospective case series study. Int J Periodontics Restorative Dent. 2022 Sep-Oct;42(5):631-637" will be used for comparison.

Study power N total: 24 Anticipated drop-out rate %: 15 Adequate power analysis and justification A power calculation before the study revealed that a sample size of 20 was necessary to detect a difference of 0.5 mm in the vertical position of the implant between planning and execution of 0.5 mm assuming a maximal standard deviation of 0.7 mm using a paired t test with 80% power and .05 level of significance.

Study intervention - test arm Study Device BLC Implant

Test treatment name Fully digital immediate placement/immediate restoration

Test Treatment description An immediate BLC implant inserted in post-extraction sites in the upper maxilla, from 15 to 25, with immediate restoration.

Primary outcome parameter Pink Esthetic Score (PES from 0 to 14), at 1 year Marginal Bone Level expressed in mm, at 1 year

Secondary outcome parameter PROMS - Patients' satisfaction using VAS scale, at day of surgery and at 1 year Duration of the procedure, at day of surgery Probing Depth (PD) and Bleeding on Probing (BoP) at 1 year

Materials and Methods Population and indication 24 adult systemically healthy patients requiring tooth extraction and single implant tooth replacement, from 1.5 to 2.5

Treatments In the case study phase, a 3D cone-beam radiograph and an intraoral scan are acquired. A computer guided surgical stent is produced from the virtual planning. By sharing the virtual planning, the laboratory designs and produces a temporary crown. On the day of surgery the tooth is extracted, the implant is inserted and the temporary is delivered. The final ceramic crown is delivered 3 months later. Follow-up will end 1 year after implant placement.

Statistical methods paired t-test

ELIGIBILITY:
Inclusion Criteria:

* adult systemically healthy patient requiring tooth extraction and single implant tooth replacement, from 1.5 to 2.5

Exclusion Criteria:

* patients not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 24 adults systemically healthy patient requiring tooth extraction and single implant tooth replacement, from 1.5 to 2.5
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score | 1 year
Marginal Bone Level | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Studio Dottor Cardaropoli, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, De Maria A. Clinical and Radiologic Evaluation of a Fully Tapered Implant with Immediate Placement in the Esthetic Zone: A Prospective Case Series Study. Int J Periodontics Restorative Dent. 2022 Sep-Oct;42(5):631-637. doi: 10.11607/prd.5682. PMID 36044694